CLINICAL TRIAL: NCT03231995
Title: Prospective Multicentre Study to Determine Respiratory Microbiome Biomarkers for the Prognostic of Clinical Course of Influenza in Children
Brief Title: Biomarkers for the Prognosis of Influenza in Children
Acronym: BMIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0175; 2017-A03035-48 (Other: IDRCB)
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Influenza
Keywords: Severe influenza; biomarkers; respiratory microbiome; prognosis
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory microbiome biomarkers (Experimental)
  Interventions: Biological: Collection of nasopharyngeal specimen collected at D0, D1, D2 and D5.

INTERVENTIONS:
Biological: Collection of nasopharyngeal specimen collected at D0, D1, D2 and D5. — Analyses will be performed on nasopharyngeal specimen collected at D0, D1, D2 and D5.
  Definition and validation of nasopharyngeal microbiome biomarkers (bacterial, viral, transcriptomic signature)

SUMMARY:
Context: Seasonal influenza affects 2.5 to 3 million people each year in France, resulting in 1500 to 2000 severe cases seen in intensive care units. The severity of influenza is related to, among other things, its respiratory or neurological complications, observed especially in children. Early determination of the severity of influenza is a critical step to avoid in appropriate treatment and care for patients and to improve their survival. Viral, human but also environmental factors have been described as having an important role in determining this severity. Several studies suggest that the nasopharyngeal microbiome may be involved in the incidence and severity of respiratory viral infections. During influenza infection, the respiratory microbiota is significantly altered. In animal models, particularly murine models, the microbiota regulates the immune response to influenza virus infection. In a retrospective preliminary study, the investigators showed that the composition of the nasopharyngeal bacterial microbiota is different between children who develop a severe or moderate influenza. This difference was observed on respiratory specimens at admission to pediatric emergencies within two days of onset of symptoms.

Hypotheses :

* The respiratory microbiome is a determining factor in the clinical course of influenza infection (benign vs. severe with respiratory or neurological complication)
* The respiratory microbiome can be used as a prognostic biomarker of the clinical course of influenza Originality: There are currently no clinical and / or virological markers to predict the clinical course of influenza infection. This study will define biomarkers of the respiratory microbiome to discriminate patients who will develop a severe influenza from those who will develop a moderate influenza. These prognostic biomarkers could be used to rapidly refer patients at risk to intensive care units, thus improving patient management and care. Moreover, at the fundamental level, this study will specify the role of the microbiome in the severity of influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Age < 5 years
* Seen in an emergency department with influenza confirmed by a positive test (polumerase chain reaction, rapide antigen detection test).

Exclusion Criteria:

* Presence of associated significant comorbidity (chronic respiratory, cardiac, neurological or metabolic pathology, prematurity, known immunodeficiency)
* Documented non-respiratory bacterial infection
* No consent
* Patient not affiliated to a national health cover

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Definition and evaluation of a microbial signature discriminating patients developing severe influenza from those developing moderate influenza | Day 30
  On nasopharyngeal specimen collected at inclusion, a microbial signature will be defined as a limited number of bacterial genomic groups (OTU Operational Taxonomic Unit), that will help discriminate the 2 groups of patients (evolution toward a severe or a moderate influenza, evaluated at hospital discharge).

SECONDARY OUTCOMES:
sequencing the hypervariable regions of the 16S RNA on the longitudinal respiratory specimens | Day 1
  We will analyze the different dynamics of the composition of the microbiome associated with different influenza evolutions. The qualitative and quantitative evolution of the microbial species present in the respiratory specimens will be evaluated by sequencing the hypervariable regions of the 16S RNA on the longitudinal respiratory specimens performed on Day 1.
sequencing the hypervariable regions of the 16S RNA on the longitudinal respiratory specimens | Day 2
  We will analyze the different dynamics of the composition of the microbiome associated with different influenza evolutions. The qualitative and quantitative evolution of the microbial species present in the respiratory specimens will be evaluated by sequencing the hypervariable regions of the 16S RNA on the longitudinal respiratory specimens performed on day 2
sequencing the hypervariable regions of the 16S RNA on the longitudinal respiratory specimens | Day 5
  We will analyze the different dynamics of the composition of the microbiome associated with different influenza evolutions. The qualitative and quantitative evolution of the microbial species present in the respiratory specimens will be evaluated by sequencing the hypervariable regions of the 16S RNA on the longitudinal respiratory specimens performed on day 5

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CIC groupement Hospitalier Est - Hospices Civils de Lyon, Lyon
  - Hopital Nord, Saint-Etienne